CLINICAL TRIAL: NCT02133430
Title: Optimized Anesthesia to Reduce Incidence of Postoperative Delirium in Elderly Undergoing Elective, Non-cardiac Surgery: a Randomized Controlled Trial (POD-II)
Brief Title: Optimized Anesthesia to Reduce Incidence of Postoperative Delirium
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Dr. Yodying Punjasawadwong, MD, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ANE-2556-01778
Record Dates: First submitted 2014-05-02; First posted 2014-05-08 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bispectral index (BIS) group (Experimental): Bispectral index as measured by a BIS Processor is used to guide doses of anesthetic for maintaining the BIS values of 40-60
  Interventions: Device: Bispectral index, as measured by a BIS processor
- Control group (No Intervention): Clinical signs is used to guide doses of anestheitics.

INTERVENTIONS:
Device: Bispectral index, as measured by a BIS processor — Comparisons of incidence of postoperative delirium.
  Other Names: BIS PROCESSOR, MODEL QE-910P, NIHON KOHDEN CORPORATION
  Arms: Bispectral index (BIS) group

SUMMARY:
The purpose of this study is to compare the difference of incidence of postoperative delirium between patients received general anesthesia guided by Bispectral index (BIS) and patients received general anesthesia using standard technique.

DETAILED DESCRIPTION:
General anesthesia is one of precipitating factor of postoperative delirium which Its mechanism is still unknown. General anesthesia can affect on pattern of electroencephalograph. Previous studies showed that patients received BIS guided anesthesia could wake up faster, earlier extubation and stay in recovery room shorter compared to standard general anesthesia. Optimized level of anesthesia by BIS could reduce cognitive dysfunction in elderly patients and reduce biological marker of brain injury. Therefore, the investigators hypothesized that adjustment of general anesthesia by BIS guided could protect central nervous system and reduce incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients age equal or more than 65 years.
* Patients undergoing general anesthesia.
* Patients undergoing scheduled, non-cardiac surgery

Exclusion Criteria:

* Patients undergoing neurosurgery.
* Patients cannot understand Thai language.
* Patients who have severe visual or hearing impairment.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients have postoperative delirium | Participants will be followed during the duration of hospital stay, an expected avarage of two weeks.
  Assess postoperative delirium by using Confusion Assessment Method for intensive care unit (CAM-ICU) at recovery room and Confusion Assessment Method at inpatient ward.

SECONDARY OUTCOMES:
Number of patients with impaired cognitive function | Up to 6 months
  Assessed postoperative cognitive function by using Mini-Mental State Examination and Montreal Cognitive Assessment (MoCA) .
Time to recovery | The end of surgery
  Time between end of anesthesia and eye opening, spontaneous breathing, and extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yodying Punjasawadwong, MD, Principal Investigator — Department of Anesthesiology, Faculty ofMedicine, Chiang Mai, University, Chiang Mai, Thailand; Dr. Tanyong Pipanmekaporn, MD, Study Director — Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand,50200
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Maung, Chiang Mai, Thailand

REFERENCES:
- See also: Sponsor's website — http://www.med.cmu.ac.th